CLINICAL TRIAL: NCT05458934
Title: Analysis of Exhaled Breath From Patients With Lung-/Airway Diseases (BigExBrESs)
Acronym: BigExBrESs
Status: Recruiting | Type: Observational
Sponsor: University of Zurich (Other)
Collaborators: Deep Breath Intelligence (DBI) (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2021-00539
Record Dates: First submitted 2022-06-30; First posted 2022-07-14 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Lung-/Airway Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lung-/Airway diseases: Patients with lung-/airway diseases
  Interventions: Other: No intervention
- Controls: Participants without lung-/airway disease
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — no intervention

SUMMARY:
Ananlyis of exhaled breath of patients with lung-/airway diseases to identify and distinguish respiratory diseases, and improve the disease manangament.

DETAILED DESCRIPTION:
Breath analysis offers a unique opportunity to non-invasively retrieve unlimited samples of relevant information on the ongoing internal biochemical processes, as parts of the most volatile components in blood reach the gas phase and are subsequently exhaled (e.g. detection of ethanol in breath). Analysis of exhaled breath provides biochemical information about the metabolism and the pathophysiological state. Chemical analysis of exhaled breath with mass spectrometry identified numerous volatile organic compounds (VOCs) [low molecular weightcomponents:< 500 Dalton (Da)]. Using Big Data analytics, specific patterns of diverse respiratory disease (e.g. for COPD and asthma) can be identified and the different diseases can be distinguished from each other. Specific Big Data Analytics might also improve the management of disease (e.g.avoiding of exacerbations) by identifying early signs of exacerbation risk.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age ≥ 18 years at study entry

Exclusion Criteria:

* Physical or intellectual impairment precluding informed consent or protocol adherence
* Known pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: General population
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2021-05-11 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Molecular breath pattern | at baseline
  Comparison of molecular weights of breath features from patients with different respiratory diseases

SECONDARY OUTCOMES:
Change in molecular breath pattern | over one year
  Change in the molecular breath pattern during the course of the disease (untargeted approach)
Symptoms | at baseline
  Correlation/Association of molecular weights of specific breath features with symptoms (e.g. dyspnea)
Inflammatory markers | at baseline
  Correlation/Association of molecular weights of specific breath features with inflammatory markers (e.g. eosinophils)
Controls | at baseline
  Differentiation of molecular breath pattern (m/z ratios of molecules in exhaled breath) between diseased patients and participants without respiratory disease (untargeted approach)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
if requested

REFERENCES:
- [Derived] Basler S, Fricke K, Sievi NA, Arvaji A, Schmidt F, Herth J, Baur DM, Kohler M, Ulrich S, Lichtblau M. Exploring breath metabolomics as a non-invasive tool for detecting pulmonary vascular disease. Eur Heart J Open. 2025 May 23;5(3):oeaf060. doi: 10.1093/ehjopen/oeaf060. eCollection 2025 May. PMID 40474893